CLINICAL TRIAL: NCT07184346
Title: Comparison of Conventional, Digital, and Optical Jaw Tracking Techniques for Recording Centric Relation: An Evaluation of Accuracy
Brief Title: Accuracy of Centric Relation Recording: Conventional to Optical
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mohammed Bin Rashid University of Medicine and Health Sciences (Other)
Responsible Party: Principal Investigator, Haitham Elbishari, Associate Professor, Mohammed Bin Rashid University of Medicine and Health Sciences
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: MBRU-HBMCDM-RG2024-05
Record Dates: First submitted 2025-05-03; First posted 2025-09-19 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Centric Relation Registration

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Accuracy of Centric Relation Record (Control) (Experimental): Centric relation will be recorded using a conventional method with a 2 mm Kois deprogrammer and polyvinyl siloxane (PVS) bite registration. Alginate impressions and facebow records will be taken, mounted on a semi-adjustable articulator, and digitized with a laboratory scanner.
  Interventions: Other: Control
- Accuracy of Centric Relation record IOS (Experimental): Centric relation will be recorded using an intraoral scanner. Maxillary and mandibular arches will be scanned, and the Kois deprogrammer with PVS registration will be used to digitally capture mandibular position
  Interventions: Device: Intra Oral Scanner
- Accuracy of Centric Relation record ModJaw (Experimental): Centric relation will be recorded using the ModJaw optical jaw tracking system (4D jaw tracker). Previously acquired scans will be imported into ModJaw, and the kois deprogrammer will standardize mandibular position during registration
  Interventions: Device: Mod Jaw

INTERVENTIONS:
Other: Control — Control Group
  Arms: Accuracy of Centric Relation Record (Control)
Device: Intra Oral Scanner — Experimental group 1
  Arms: Accuracy of Centric Relation record IOS
Device: Mod Jaw — 4 D Jaw Tracker
  Arms: Accuracy of Centric Relation record ModJaw

SUMMARY:
The current study aims to evaluate the accuracy of different techniques used to record the centric relation.

The sample size was determined based on a previous study by Revilla-León et al. (2023), which indicated that 18 participants per group would provide sufficient power for statistical analysis. Eligible participants will be adults above 18 years of age with good oral health who are fully or partially dentate. Exclusion criteria include complete edentulism, absence of posterior stops, temporomandibular joint disorders, and limited mouth opening.

Centric relation (CR) will be recorded for all participants using three methods. In Group 1 (Conventional), a 2 mm Lucia jig fabricated from pattern resin (Dura-lay) will be positioned intraorally with the participant reclined at 45°. Polyvinyl siloxane (PVS) bite registration material will be injected bilaterally from the canines to first molars and allowed to set. Alginate impressions, facebow records, and subsequent mounting on a semi-adjustable articulator will be performed, and the casts will be digitized with a laboratory scanner. In Group 2 (Intraoral Scanner), the iTero Element scanner (Align Technology, San Jose, CA) will be used to capture maxillary and mandibular arches. The same Lucia jig will be placed intraorally, and the bite will be digitally captured using the PVS record. In Group 3 (Optical Jaw Tracking), the Modjaw system will be used with previously acquired iTero scans. The Lucia jig will again standardize mandibular position during CR registration. All recordings will be performed by a single experienced prosthodontist to ensure consistency.

For accuracy assessment, STL files from all recordings will be imported into Geomagic Control X (3D Systems). Six digital markers will be placed on maxillary and mandibular reference scans at standardized anatomical landmarks (buccal surfaces of first molars, canines, and central incisors). Thirty-six baseline inter-landmark distances will be calculated. Each experimental scan will then be aligned to the reference scan using a best-fit alignment protocol, with marker coordinates transferred from the reference scan to maintain consistency and avoid manual errors. Inter-landmark distances will be recalculated for each experimental scan. Accuracy will be assessed in terms of trueness (mean absolute deviation between reference and experimental measurements) and precision (consistency of distances within each group).

Data will be statistically analyzed using analysis of variance (ANOVA), with significance set at p < 0.05.

ELIGIBILITY:
Inclusion Criteria:

1. Adults above the age of eighteen years
2. Presenting with good oral health
3. Fully or partially dentate

Exclusion Criteria:

1. Fully edentulous
2. Partially dentate with lack of posterior stops
3. Temporomandibular Joint Disorders (TMD)
4. Limited mouth opening

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-09-30 (Estimated); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Accuracy of Centric Relation Recording (Trueness and Precision in millimeters) | Baseline (Day 5, immediately after centric relation recording).
  Accuracy will be assessed by evaluating trueness and precision of centric relation (CR) records obtained with three techniques: conventional, intraoral scanner, and ModJaw optical jaw tracker. Trueness will be calculated as the mean absolute deviation (mm) between inter-landmark distances on reference STL scans and experimental scans using Geomagic Control X software. Precision will be measured as the standard deviation of repeated inter-landmark distances within each group. Data will be reported as mean ± SD values

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ries JM, Grunler C, Wichmann M, Matta RE. Three-dimensional analysis of the accuracy of conventional and completely digital interocclusal registration methods. J Prosthet Dent. 2022 Nov;128(5):994-1000. doi: 10.1016/j.prosdent.2021.03.005. Epub 2021 Apr 19. PMID 33888327
- [Background] Revilla-Leon M, Subramanian SG, Ozcan M, Krishnamurthy VR. Clinical Study of the Influence of Ambient Light Scanning Conditions on the Accuracy (Trueness and Precision) of an Intraoral Scanner. J Prosthodont. 2020 Feb;29(2):107-113. doi: 10.1111/jopr.13135. Epub 2019 Dec 30. PMID 31860144
- [Background] Renne W, Ludlow M, Fryml J, Schurch Z, Mennito A, Kessler R, Lauer A. Evaluation of the accuracy of 7 digital scanners: An in vitro analysis based on 3-dimensional comparisons. J Prosthet Dent. 2017 Jul;118(1):36-42. doi: 10.1016/j.prosdent.2016.09.024. Epub 2016 Dec 23. PMID 28024822
- See also: Related Info — http://mbru.ac.ae